CLINICAL TRIAL: NCT06357767
Title: Healing Within: Smoking Cessation Intervention for American Indian Women Experiencing Intimate Partner Violence
Brief Title: Smoking Cessation Intervention for American Indian Women Experiencing Intimate Partner Violence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Black Hills Center for American Indian Health (Other)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S06GM146079 (NIH)
Record Dates: First submitted 2024-01-16; First posted 2024-04-10 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Smoking Cessation; Cigarette Smoking
MeSH Terms: conditions — Smoking Cessation; Cigarette Smoking

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healing Within (Experimental): A culturally-tailored, trauma-informed group intervention to support smoking cessation by leveraging Lakota values, mindfulness, and a storytelling approach.
  Interventions: Behavioral: Healing Within: Smoking Cessation Intervention for American Indian Women Experiencing Intimate Partner Violence

INTERVENTIONS:
Behavioral: Healing Within: Smoking Cessation Intervention for American Indian Women Experiencing Intimate Partner Violence — A culturally-tailored, trauma-informed group intervention to support smoking cessation by leveraging Lakota values, mindfulness, and a storytelling approach.

SUMMARY:
The goal of this project is to refine and test a culturally-tailored smoking cessation intervention for American Indian women who have experienced intimate partner violence (IPV). The primary aims of this study are to: (a) use a community-based participatory approach to refine intervention materials and finalize pilot intervention methodology for a culturally tailored, trauma-informed smoking cessation intervention for AI women who have experienced IPV; (b) examine feasibility, acceptability, satisfaction, and preliminary efficacy of the intervention; and (c) explore changes in alcohol and drug use over the course of the intervention.

Participants will be asked to participate in the 8-week Healing Within: Smoking Cessation Intervention for American Indian Women Experiencing Intimate Partner Violence, and complete interviews at baseline, end-of-treatment, and three months from the end of treatment.

DETAILED DESCRIPTION:
Cigarette smoking and intimate partner violence (IPV) are preventable, major public health concerns that result in severe physical and psychological consequences. Women who have experienced IPV are more likely to suffer from substance use, depression, anxiety, and post-traumatic stress disorder --all of which are risk factors for smoking. Among women who have experienced IPV, post-traumatic stress disorder severity is related to nicotine dependence. Smoking prevalence among women who have experienced IPV is as high as 51% to 70%, which is two to three times greater than among women nationally. The high prevalence of smoking among women who have experienced IPV is a critical health concern because approximately one-third of U.S. women will experience IPV during their lifetime.

American Indian women, including Northern Plains Tribal women, experience the highest proportion of IPV among women from any racial/ethnic group. Furthermore, smoking prevalence among Northern Plains Tribal women is among the highest in the U.S. These high rates of smoking coupled with early age of initiation are accompanied by rising rates of mortality from cardiovascular disease and lung cancer, which are leading causes of death among this high risk group.

Multiple health interventions have been developed for women who have experienced IPV, including for alcohol and drug use, given the high rates of these co-occurring problems. However, there have been no smoking cessation interventions among them. While smoking cessation approaches for American Indians typically address the differences of ceremonial versus commercial tobacco, such programs have not incorporated trauma-informed strategies-a framework that understands and responds to the impact of trauma by emphasizing physical, psychological, and emotional safety. Further, mindfulness-based approaches are shown to mitigate habitual patterns of reactive or addictive behaviors by increasing awareness of reactivity and automated (e.g., smoking) behavior, allowing greater flexibility in response to cravings. These strength-based trauma-informed and mindfulness approaches are consistent with the values of American Indian culture and create opportunities for individuals who have been traumatized to rebuild a sense of choice, control, and safety. The physical health benefits to be experienced by American Indian women smokers upon quitting are significant. These include improvements in circulation and respiratory function, decreased risk of myocardial infarction and stroke, and decreased secondhand smoke exposure to family members. Additionally, the mental health benefits of a trauma-informed, mindfulness-based approach to interventions in general are clearly documented.

The research team used an interactive, highly participatory approach to collect and use qualitative data to inform the initial development of a culturally tailored, trauma-informed smoking cessation intervention for Northern Plains Tribal women who have experienced IPV. Therefore, consistent with Stage 1a and 1b of the Stage Model of intervention development, the primary objective of this application is to finalize the 8-session novel intervention and examine its feasibility, acceptability, and satisfaction.

To achieve this goal, the following Specific and Technical Aims will be addressed:

Aim 1. Use a community-based participatory approach with a Community Advisory Board to refine intervention materials (including facilitator manual and training materials) and finalize pilot intervention methodology.

Aim 2. Conduct a single arm intervention trial enrolling 48 Northern Plains Tribal women smokers who have experienced IPV to examine: a) the primary study outcomes of feasibility, acceptability, and satisfaction with the culturally tailored, trauma-informed mindfulness smoking cessation intervention and b) the secondary study outcome of quit attempts and biochemically verified smoking abstinence prevalence at 3 and 6-months follow-up, which will gauge the effectiveness of the intervention.

Exploratory Aim. Concurrently, the investigators will explore changes in drug and alcohol use given the proposed intervention's central focus on personal and historical trauma among American Indian women as contributors to addiction and consistent with a focus on poly- vs. single substance use.

Smoking cessation is among the most impactful behavior changes - it is effective in reducing morbidity and premature death. This project capitalizes on the Black Hills Center for American Indian Health's excellent and long-standing relationship with the Rapid City Indian Community, principally Lakota. Results will be among the very first evidence concerning smoking cessation efforts in this highly resilient though vulnerable and understudied population. Finally, this project's highly participatory approach will further strengthen tribal community partners' knowledge, expertise, and support for research conducted in a respectful and community-based framework. Findings will be used to inform a fully powered RCT to test this intervention in a Stage II trial.

ELIGIBILITY:
Inclusion Criteria:

* American Indian woman from the Northern Plains
* Live in Rapid City, SD or surrounding area
* Willing to quit smoking during study participation
* 18 years of age or older
* Smoking at least five cigarettes per day
* Experienced physical and/or psychological IPV in the past three months

Exclusion Criteria:

* Inability to give consent and/or adequately complete questionnaires due to cognitive impairment.
* Self-reported pregnancy or intention to become pregnant during the intervention period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only participants who self-identify as cisgender women will be included.
Enrollment: 48 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Trauma-Informed Practice Scales (TIPS) | Up to week 8
  Participants perception of cultural responsiveness of the intervention will be assessed using the 8-item Cultural Responsiveness and Inclusivity subscales of the TIPS as an index of intervention acceptability/likability. Items are rated on a 0-3 Likert scale, and mean scores are computed. Scores range from 0-3, with higher scores representing receipt of more trauma-informed, culturally responsive services.
Session Rating Scale (SRS) | Up to week 8
  Participant ratings of working alliance will be assessed using the SRS as an index of intervention acceptability/likability. The SRS is a 4-item visual analog instrument. Each item is assessed using a 0-10 point scale. A total score is computed by summing each item. Scores will range from 0-60, with an overall score of 36, or 9 on any item, indicating potential concerns in working alliance.
Group Attitude Scale (GAS) | Up to week 8
  Group cohesion will be assessed using a modified version of the GAS an an index of intervention acceptability/likability. The 20 items are rated on a 1-5 Likert scale. A total score is computed by averaging the items. Scores range from 1-5, with higher scores indicating more group cohesion.

SECONDARY OUTCOMES:
Biochemical verification of smoking status | Baseline
  Expired breath carbon monoxide will be measured using a carbon monoxide breath monitor. Carbon monoxide readings greater than 3ppm are indicative of smoking.
Biochemical verification of smoking status | End of treatment (approximately 8 weeks following baseline)
  Expired breath carbon monoxide will be measured using a carbon monoxide breath monitor. Carbon monoxide readings greater than 3ppm are indicative of smoking.
Biochemical verification of smoking status | 3-months post treatment completion
  Expired breath carbon monoxide will be measured using a carbon monoxide breath monitor. Carbon monoxide readings greater than 3ppm are indicative of smoking.
Quit Attempts | Baseline
  Lifetime quit attempts of at least 24 hours will be assessed by self-report.
Quit Attempts | End of treatment (approximately 8 weeks following baseline)
  Quit attempts of at least 24 hours will be assessed by self-report referencing the time since baseline.
Quit Attempts | 3-months post treatment completion
  Quit attempts of at least 24 hours will be assessed by self-report referencing the time since the end-of-treatment follow-up interview.

OTHER OUTCOMES:
Alcohol Use Disorders Identification Test (AUDIT) | Baseline
  The AUDIT is a 10-item self-report instrument designed to identify individuals for whom the use of alcohol places them at risk for alcohol problems or who are experiencing such problems. The AUDIT items ask about the past year, although a few items have no specific time reference. AUDIT total scores can range from 0 to 40 with higher scores indicating worse outcomes, and scores of 8 or above have been used to identify individuals who may be at risk for or who are experiencing alcohol problems. Considerable empirical evidence supports the instrument's internal consistency.
Alcohol Use Disorders Identification Test (AUDIT) | End of treatment (approximately 8 weeks following baseline)
  The AUDIT is a 10-item self-report instrument designed to identify individuals for whom the use of alcohol places them at risk for alcohol problems or who are experiencing such problems. The AUDIT items ask about the past year, although a few items have no specific time reference. AUDIT total scores can range from 0 to 40 with higher scores indicating worse outcomes, and scores of 8 or above have been used to identify individuals who may be at risk for or who are experiencing alcohol problems. Considerable empirical evidence supports the instrument's internal consistency.
Alcohol Use Disorders Identification Test (AUDIT) | 3-months post treatment completion
  The AUDIT is a 10-item self-report instrument designed to identify individuals for whom the use of alcohol places them at risk for alcohol problems or who are experiencing such problems. The AUDIT items ask about the past year, although a few items have no specific time reference. AUDIT total scores can range from 0 to 40 with higher scores indicating worse outcomes, and scores of 8 or above have been used to identify individuals who may be at risk for or who are experiencing alcohol problems. Considerable empirical evidence supports the instrument's internal consistency.
NIDA ASSIST | Baseline
  The NIDA ASSIST is a validated screening tool recommended to assess level of risk related to substance use.
NIDA ASSIST | End of treatment (approximately 8 weeks following baseline)
  The NIDA ASSIST is a validated screening tool recommended to assess level of risk related to substance use.
NIDA ASSIST | 3-months post treatment completion
  The NIDA ASSIST is a validated screening tool recommended to assess level of risk related to substance use.

CONTACTS AND LOCATIONS:
Locations (1):
- Black Hills Center for American Indian Health, Rapid City, South Dakota, United States